CLINICAL TRIAL: NCT02058745
Title: SmartCare: Innovations in Caregiving Interventions
Acronym: SmartCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Paula Sherwood, Professor, Vice Chair of Research, Dept. of Acute and Tertiary Care, School of Nursing; Professor, Dept. of Neurological Surgery, School of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO11060487; R01NR013170 (NIH)
Record Dates: First submitted 2013-11-19; First posted 2014-02-10 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Primary Malignant Brain Tumors
Keywords: Neuro-oncology; Caregivers; Intervention Research; Representational Approach; Cognitive Behavioral Therapy; Family; Internet
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CAU+ (Enhanced Care as Usual) (Active Comparator): CAU+ (Enhanced Care as Usual) is defined as the care received from the care recipient's oncologist supplemented by unlimited access to three components of the study website: caregiver guides, links to web-based resources, and a basic friends and family page for the 10 month duration of the study.
  Interventions: Behavioral: CAU+ (Enhanced Care as Usual)
- CAU+ and SmartCare (Experimental): CAU+ (Enhanced Care as Usual) for eight weeks, followed by eight weeks of SmartCare. SmartCare is a web-based, nurse guided intervention for caregivers based on the Representational Approach of symptom management.
  Interventions: Behavioral: CAU+ (Enhanced Care as Usual); Behavioral: SmartCare
- CAU+ and Beating the Blues and SmartCare (Experimental): CAU+ (Enhanced Care as Usual) and Beating the Blues concurrently for eight weeks, followed by SmartCare for eight weeks. Beating the Blues is an established, web-based, self-directed, cognitive behavioral therapy for managing depressive symptoms.
  Interventions: Behavioral: CAU+ (Enhanced Care as Usual); Behavioral: Beating the Blues; Behavioral: SmartCare

INTERVENTIONS:
Behavioral: CAU+ (Enhanced Care as Usual) — CAU+ is defined as the care received from the care recipient's oncologist supplemented by unlimited access to three components of the study website: caregiver guides, links to web-based resources, and a basic friends and family page. These resources are routinely available on the Internet. We provide these as a "one-stop shopping" resource in order to standardize care as usual for caregivers. All caregivers will be sent personalized e-mails from the project director every week during the intervention period.
Behavioral: Beating the Blues — Beating the Blues is an established, self-directed, web-based cognitive behavioral therapy program for managing depressive symptoms. Caregivers are asked to complete 8 weekly sessions, each lasting approximately 50 minutes. Participants are also given simple "homework" after each lesson.
  Arms: CAU+ and Beating the Blues and SmartCare
Behavioral: SmartCare — SmartCare is a web-based, nurse guided intervention for caregivers based on the Representational Approach of symptom management. The RA builds on traditional cognitive-behavioral interventions by promoting in depth reflection of previous and current experiences, beliefs, and knowledge (referred to as representations) prior to providing new information or engaging in problem-solving.
  Arms: CAU+ and Beating the Blues and SmartCare; CAU+ and SmartCare

SUMMARY:
This is a study to evaluate the effectiveness of using an established intervention for depressive symptom management in conjunction with a needs-based caregiver intervention for improving the psychological and physical health of family caregivers of persons recently diagnosed with a Primary Malignant Brain Tumor.

DETAILED DESCRIPTION:
We have designed a needs-based intervention to improve neuro-oncology caregivers' health. Our novel approach treats depressive symptoms prior to implementing a needs-based intervention in a sample of PMBT family caregivers who score above threshold on depressive symptoms. Study outcomes are psychological responses (unmet needs, depressive symptoms, anxiety, and burden) and physical responses (levels of stimulated and circulating IL-6 and IL-1β, C-reactive protein, peripheral blood mono-nuclear cells, physical symptoms, and new diagnoses or exacerbations of co-morbid conditions). The proposed study addresses research priorities set by both NCI and NINR to improve the quality of life of patients and their families and NINR's emphasis on integrating bio-behavioral science and adopting, adapting and generating new technologies.

Primary aims:

1. Compare the efficacy of a) an intervention for depressive symptoms (Beating the Blues) delivered prior to a needs-based caregiver intervention (SmartCare©) versus b) SmartCare© alone versus c) enhanced care as usual (CAU+) in improving caregivers' psychological and physical responses.

   H1: At 4- and 6-months, caregivers who receive Beating the Blues prior to SmartCare© will display improved psychological and physical responses compared to caregivers who receive CAU+.

   H2: At 4- and 6-months, caregivers who receive SmartCare© alone will display improved psychological and physical responses compared to caregivers who receive CAU+.

   H3: At 4- and 6-months, caregivers who receive Beating the Blues prior to SmartCare© will display improved psychological and physical responses compared to those who receive SmartCare© alone.
2. Compare the efficacy of Beating the Blues versus CAU+ in improving subjects' short-term psychological and physical responses.

H1: At 2-months following baseline, caregivers who receive Beating the Blues will display improved psychological and physical responses compared to CAU+.

Exploratory aims:

1. Determine whether any changes in psychological and physical health resulting from receiving Beating the Blues prior to SmartCare© or SmartCare© alone are maintained at 10-months after baseline.
2. Evaluate whether the effect of Beating the Blues + SmartCare© (vs. SmartCare© alone) on 4- and 6-month psychological and physical responses is mediated by 0- to 2-month changes in depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

Care recipient:

* Over 21 years of age.
* Newly (within 1 month) diagnosed with a PMBT (tumor verified via pathology report to be a glioblastoma multiforme, anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic oligoastrocytoma, medulloblastoma, or anaplastic ependymoma).

Caregiver:

* Primary nonprofessional, non-paid caregiver, as identified by the care recipient.
* Over 21 years of age with telephone access.
* Reads-speaks English
* Obtains a score of >6 on the shortened CES-D.
* Caregivers may or may not be receiving pharmacotherapy for depressive symptoms

Exclusion Criteria:

Caregiver:

* Currently considers self to be a primary caregiver for anyone else other than children
* Currently receiving any type of formal counselling for depressive symptoms

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2017-06-14 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
Change in depression from baseline at 4 months on the shortened CES-D | Baseline and 4 months
  Depressive symptoms will be measured using the 10-item shortened version of the Center for Epidemiologic Studies - Depression (CES-D).

SECONDARY OUTCOMES:
Change in unmet needs from baseline at 4 months on the CNS | Baseline and 4 months
  Unmet Needs will be measured via the Caregiver Needs Screen (CNS) questionnaire.
Change in mastery from baseline at 4 months on the Caregiver Mastery Scale | Baseline and 4 months
  Mastery will be measured using the Caregiver Mastery Scale.
Change in optimism from baseline at 4 months on the Life Orientation Test | Baseline and 4 months
  Optimism will be measured using the Life Orientation Test.
Change spirituality from baseline at 4 months on the FACIT. | Baseline and 4 months.
  Spirituality will measured using the Functional Assessment of Chronic Illness Therapy - Sp (FACIT).
Change in oversight demand from baseline at 4 months on the caregiver vigilance scale. | Baseline and 4 months
  Caregiver oversight demand will be measured using the four item Caregiver Vigilance Scale.
Change in social support from baseline at 4 months on the ISEL. | Baseline and 4 months.
  Social support will be measured using the Interpersonal Support Evaluation List (ISEL). Subjects rate the availability of three types of social support (appraisal, belonging, and tangible).
Change in occupational functioning from baseline at 4 months on the WLQ. | Baseline and 4 months.
  Caregiver occupational functioning will be measured by general questions related to employment status and the Work Limitations Questionnaire (WLQ).
Changes in positive aspects of providing care from baseline at 4 months on the PAC. | Baseline and 4 months
  Positive aspects of providing care will be measured using the Positive Aspects of Caregiving (PAC) scale.
Change in unmet needs from baseline at 6 months on the CNS | Baseline and 6 months
  Unmet Needs will be measured via the Caregiver Needs Screen (CNS) questionnaire.
Change in mastery from baseline at 6 months on the Caregiver Mastery Scale | Baseline and 6 months
  Mastery will be measured using the Caregiver Mastery Scale.
Change in optimism from baseline at 6 months on the Life Orientation Test | Baseline and 6 months
  Optimism will be measured using the Life Orientation Test.
Change spirituality from baseline at 6 months on the FACIT. | Baseline and 6 months.
  Spirituality will measured using the Functional Assessment of Chronic Illness Therapy - Sp (FACIT).
Change in oversight demand from baseline at 6 months on the caregiver vigilance scale. | Baseline and 6 months
  Caregiver oversight demand will be measured using the four item Caregiver Vigilance Scale.
Change in social support from baseline at 6 months on the ISEL. | Baseline and 6 months.
  Social support will be measured using the Interpersonal Support Evaluation List (ISEL). Subjects rate the availability of three types of social support (appraisal, belonging, and tangible).
Change in occupational functioning from baseline at 6 months on the WLQ. | Baseline and 6 months.
  Caregiver occupational functioning will be measured by general questions related to employment status and the Work Limitations Questionnaire (WLQ).
Changes in positive aspects of providing care from baseline at 6 months on the PAC. | Baseline and 6 months
  Positive aspects of providing care will be measured using the Positive Aspects of Caregiving (PAC) scale.

CONTACTS AND LOCATIONS:
Overall Officials: Paula R Sherwood, PhD, Principal Investigator — University of Pittsburgh, School of Nursing; Heidi S Donovan, PhD, Principal Investigator — University of Pittsburgh, School of Nursing
Locations (1):
- University of Pittsburgh, School of Nursing, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable data will be shared with interested parties in agreement with University policy.

REFERENCES:
- [Derived] Sherwood PR, Boele F, Weimer J, Marsland A, Drappatz J, Armstrong TS, Terhorst L, Donovan HS. Neuro-oncology Caregiver Intervention Associated With Changes in C-Reactive Protein. Cancer Nurs. 2025 Apr 22. doi: 10.1097/NCC.0000000000001507. Online ahead of print. PMID 40266659
- [Derived] Boele FW, Weimer JM, Marsland AL, Armstrong TS, Given CW, Drappatz J, Donovan HS, Sherwood PR. The effects of SmartCare(c) on neuro-oncology family caregivers' distress: a randomized controlled trial. Support Care Cancer. 2022 Mar;30(3):2059-2068. doi: 10.1007/s00520-021-06555-5. Epub 2021 Oct 16. PMID 34655326
- [Derived] Boele FW, Weimer J, Zamanipoor Najafabadi AH, Murray L, Given CW, Given BA, Donovan HS, Drappatz J, Lieberman FS, Sherwood PR. The Added Value of Family Caregivers' Level of Mastery in Predicting Survival of Glioblastoma Patients: A Validation Study. Cancer Nurs. 2022 Sep-Oct 01;45(5):363-368. doi: 10.1097/NCC.0000000000001027. Epub 2021 Sep 30. PMID 34608049